CLINICAL TRIAL: NCT03461419
Title: Use of Cellular Stromal Vascular Fraction in Multiple Sclerosis
Brief Title: Use of Stromal Vascular Fraction in Multiple Sclerosis
Acronym: GARM-MS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn [COVID restrictions prevent patient enrollment or treatment. Clinical Trial facility is being closed due to viral limitations and loss of staff to perform]
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Global Alliance for Regenerative Medicine (Other)
Responsible Party: Principal Investigator, Robert W. Alexander, MD, FICS, Prinicipal Investigator, Healeon Medical Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GARM-MS
Record Dates: First submitted 2018-01-23; First posted 2018-03-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis; Autoimmune
Keywords: Multiple Sclerosis; Demyelinating Disease; Nervous System Degenerative Disease; Autoimmune Disease
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Microcannula Harvest Adipose Stroma (Experimental): Acquisition of AD-tSVF via closed syringe microcannula
  Interventions: Procedure: Microcannula Harvest Adipose Stroma
- Centricyte 1000 (Experimental): Autologous Adipose-Derived Tissue Stromal Vascular Fraction (AD-tSVF) via enzymatic isolation/concentration closed system to create cellular stromal vascular fraction (cSVF)
  Interventions: Device: Centricyte 1000
- Sterile Normal Saline IV (Experimental): Re-suspension of cSVF pellet in Sterile Normal Saline Intravenous Delivery
  Interventions: Procedure: Sterile Normal Saline IV Deployment of cSVF

INTERVENTIONS:
Procedure: Microcannula Harvest Adipose Stroma — Use of Disposable, Closed Syringe Microcannula Harvest Autologous Adipose Stroma and Stem/Stromal Cells
  Arms: Microcannula Harvest Adipose Stroma
Device: Centricyte 1000 — Centricyte 1000 closed system digestion of stromal vascular fraction to isolate and concentrate stem/stromal cells associated with microvasculature
  Arms: Centricyte 1000
Procedure: Sterile Normal Saline IV Deployment of cSVF — Sterile Normal Saline Suspension cSVF in 500 cc for Intravenous Delivery Including 150 micron in-line filtration
  Arms: Sterile Normal Saline IV

SUMMARY:
Purpose of study is to determine safety and efficacy of use of autologous Adipose-Derived cellular Stromal Vascular Fraction (AD-cSVF) suspended in Normal Saline and delivered via intravascular system of quality of life and alteration of documented Advanced Muscular Sclerosis (MS). It is believed that the heterogeneous cell population which includes multipotent stem/stromal cells plus non-multipotent cellular elements are capable of immune modulation/inflammatory modulation properties. Exam of disease progression and quality of life changes will be evaluated by sophisticated mathematical non-biased MRI analysis.

DETAILED DESCRIPTION:
Advanced Multiple Sclerosis (MS), defined as a non-medication responsive MS, which is a demyelination disease which features damage to insulating covers of nerve cells in the brain and spinal cord. This damage or degenerative changes disrupts the ability of parts of the nervous system to communicate, resulting in range of signs and symptoms which include physical and mental changes.

Symptoms are variable and often include visual changes, sensory irregularities, and motor coordination. MS has several forms which result in new symptoms in either isolated attacks (relapsing forms) or gradual increasing symptoms (progressive forms). In most cases, severe side effects or non-responsive cases to traditional MS medications on the market, have not proven to be acceptable, totally safe (without severe side effects) or clinically efficacious.

While cause is not clear, mechanisms have been suggested association with loss of the immune system or failure to produce myelin-producing cells. Some suggest a genetic predisposition or environmental factor, but the exact causation in all cases have not been elucidated.

Medications have been developed, but remain modestly effective and possessing major side effects and poorly tolerated. Alternative treatments, including physical therapy and some stem/stromal therapies have become more common.

Three main characteristics of MS are: 1). Lesion formations in the central nervous system (called Plaques); 2). Inflammation; 3). Destruction of myelin sheaths of neurons. This demyelination is thought to stimulate the inflammatory processes due to action of a lymphocyte group known at T-cell which seems to recognize patient's own myelin as foreign and proceeds to attack it (known as "autoreactive lymphocytes").

Traditionally, exacerbation's are often treated with high dose intravenous steroids which may be of short term reduction of symptoms, not addressing the underlying causation. Current medications available for treatment are expensive and fraught with major side effects, making their use very difficult and producing limited measured value.

With the advent of convenient adipose harvesting and processing in closed systems, the ability to easily and safely acquire significant of stem/stromal cells, studies are underway to utilize autologous stem/stromal cells. This study is aimed at evaluation of the safety profile (adverse reactions & severe adverse reaction) of the closed syringe, microcannula harvesting of subdermal fat deposits. This autologous cell group obtained with isolation and concentration of cells within the stromal vascular fraction (SVF) via enzymatic digestion, and deployed via intravascular routes. As these cells are very small, there is belief that they are able to pass into the cerebral fluids in defects of the blood brain barrier (BBB) or are small enough to pass into the fluids of the CNS (central nervous system).

Recent availability of a highly complex analytic program will be used to assess changes in the location, numbers, volumes, demyelination of brain lesions examined by MRI (with and without contrast). This is done as a comparative analysis at intervals of baseline to 6 month minimum, and annually as available for tracking of central nervous system (CNS) changes over time and correlated with clinical progressions.

ELIGIBILITY:
Inclusion Criteria:

* Documented functional damage to central or peripheral nervous system unlikely to improve with present standard of care
* At least 6 months after onset of disease process
* If under current medical therapy (drug or surgical) for the condition, patient considered stable on that treatment and unlikely to have significant reversal of associated neurological functions damage as a result of ongoing treatments
* In estimation of providers and neurologists have the potential for improvement with AD-cSVF treatment, and be at minimal risk of potential harm from the procedure
* Over 18 year old, and capable of providing informed consent
* Medically stable and cleared by primary care physician, neurologist, or licensed practitioner that patient is felt to be reasonably expected to be expected to undergo procedures without known significant risk to health

Exclusion Criteria:

* Patient must be capable of an adequate neurologic examination and evaluation to document the pathology and ability to cooperate with examination
* Patient must be capable and willing to undergo follow up neurologic exams with investigators or their own neurologists
* Patient must be capable and competent to provide informed consent to participation
* In estimation of investigators, the patient may be at increased or significant risk of harm to the patient's general health or neurologic functions for collection of AD-cSVF collection
* Patients not medically stable, or who may be at significant risk to their health undergoing any and all procedures will not be eligible
* Women of childbearing age must not be pregnant at the time of treatment, and should refrain from becoming pregnant for 3 months post-treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events [Time Frame: Outcome measures evaluated at baseline and reviewed at 6 month intervals for average time frame of 5 years] | 6 month intervals for up to 5 years
  Activities of Daily Living (ADL)

SECONDARY OUTCOMES:
Deficits of Neurologic Functioning prior to treatment | 6 month intervals for up to 5 years
  Deficits of neurologic function identified by patient as impaired prior to treatment assessed. Examples: neurologic function may include speech, balance, motor/sensory actions, hearing, gait, strength, pain, paresthesias
Quality of Life | 6 month
  Change from baseline in general quality of life (QoL) using Health status questionnaire (Doc-25)
Brain Lesions | 6 month interval minimum for up to 5 years
  PIXYL software analysis change from baseline MRI with and without contrast; This is an objective standardized metric for analysis of demyelination, plaque formation, changes of number/volume and lessening or worsening of either data point. This is done at six month and one year minimum with option to do annually for up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Glenn C Terry, MD, Principal Investigator — GARM International
Locations (2):
- Robert W. Alexander, MD, FICS, LLC, Stevensville, Montana, United States
- Global Alliance of Regenerative Medicine (GARM) International, Roatán, Hn, Honduras

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsang BK, Macdonell R. Multiple sclerosis- diagnosis, management and prognosis. Aust Fam Physician. 2011 Dec;40(12):948-55. PMID 22146321
- [Background] Huntley A. A review of the evidence for efficacy of complementary and alternative medicines in MS. Int MS J. 2006 Jan;13(1):5-12, 4. PMID 16420779
- [Background] Hassan-Smith G, Douglas MR. Management and prognosis of multiple sclerosis. Br J Hosp Med (Lond). 2011 Nov;72(11):M174-6. doi: 10.12968/hmed.2011.72.sup11.m174. PMID 22082979
- [Background] Olsen SA. A review of complementary and alternative medicine (CAM) by people with multiple sclerosis. Occup Ther Int. 2009;16(1):57-70. doi: 10.1002/oti.266. PMID 19222053
- [Background] Luessi F, Siffrin V, Zipp F. Neurodegeneration in multiple sclerosis: novel treatment strategies. Expert Rev Neurother. 2012 Sep;12(9):1061-76; quiz 1077. doi: 10.1586/ern.12.59. PMID 23039386
- [Background] Alexander RW. Use of PIXYL software analysis of brain MRI (with & without contrast) as valuable metric in clinical trial tracking in study of multiple sclerosis (MS) and related neurodegenerative processes. Clin Trials Degener Dis 2017;2(1):1-10.